CLINICAL TRIAL: NCT05764499
Title: Physiotherapy Scoliosis Specific Exercise Improves Truncal Shift in Idiopathic Scoliosis: a 24 Month Follow up
Brief Title: Physiotherapy Scoliosis Specific Exercise Improves Truncal Shift in Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Scoliosis SOS Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ScoliosisSOS1
Record Dates: First submitted 2023-02-07; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Scoliosis; Apical Deviation; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Patients under the age of 18
  Interventions: Other: Physiotherapy Scoliosis Specific Exercise (PSSE)
- Adults: Patients 18 years old and above
  Interventions: Other: Physiotherapy Scoliosis Specific Exercise (PSSE)

INTERVENTIONS:
Other: Physiotherapy Scoliosis Specific Exercise (PSSE) — Patients completed 120 hours of group based PSSE over a four week time frame. Monday - Friday, 10.00-17.00.

SUMMARY:
Introduction: Truncal shift caused by scoliosis can be measured with a Formetric Scanner using the Maximal Thoracic Apical Deviation (MTAD) measurement. It is a well-documented complaint with regards to body-image in patients with idiopathic scoliosis (IS). Furthermore, thoracic apical deviation is an important measure in pre-operative assessment and post-operative outcomes.

Objective: The aim of this retrospective cohort study was to determine the long-term effects of an intensive course of Physiotherapy Scoliosis Specific Exercise (PSSE) on MTAD in patients with IS.

Methods: Consecutive IS patients with a single right-sided thoracic curvature who completed an intensive 4-week course of PSSE were recruited. Data was collected between April 2019 and December 2021. All patients were routinely scanned using a Formetric Scanner pre-, immediately post-, 12- and 24-months post-treatment. MTAD, measured in millimetres, was documented. Adults (>17 years old) (group 1) and children (group 2) were analysed separately.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the group treatment program in its entirety. Patients who have measurements obtained from all necessary time points. Patient who have Scoliosis and who have a primary thoracic curvature.

Exclusion Criteria:

* Patient who did not complete treatment or all measurements obtained. Patients who underwent surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were all consecutive patients at the Scoliosis SOS Clinic in London, a private healthcare clinic specializing in non-invasive treatment for Scoliosis. All patients were routinely completing their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Maximal Thoracic Apical Deviation | Pre-Treatment (Day 1 of treatment), Day 20 of treatment after study completion, an average of four weeks later, 12 months after Post-Treatment, and 24 months after Post-Treatment
  Maximal Apical Deviation measurement in mm, obtained from the DIERS 4D Formetric Scanner

SECONDARY OUTCOMES:
Body Image Score | Pre-Treatment (Day 1 of treatment), Day 20 of treatment after study completion, an average of four weeks later, 12 months after Post-Treatment, and 24 months after Post-Treatment
  Average Body Image Score. Average score from 5 categories, scored from 1-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Scoliosis SOS Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No patient information or databases will be shared outside of the clinic